CLINICAL TRIAL: NCT07148856
Title: Effect of a Combination of Myofascial Release Technique to Conventional Physiotherapy Program on Functional Outcomes in Pediatric Cerebral Palsy Post Achilles Tendon Surgery in the Gaza Strip
Brief Title: Myofascial Release Plus Physiotherapy for Children With Cerebral Palsy Post Achilles Tendon Surgery in Gaza (MFR-CP25)
Acronym: MFR-CP25
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ismail K. Al-Qudra (Other)
Responsible Party: Sponsor-Investigator, Ismail K. Al-Qudra, MSc Candidate in Orthopedic Physical Therapy, Al-Azhar University - Gaza
Organization: Al-Azhar University - Gaza (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MScPT_CP_MFR2025
Record Dates: First submitted 2025-08-23; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Cerebral Palsy Achilles Tendon Contracture Achilles Tendon Surgery
Keywords: Myofascial Release Physiotherapy Physical Therapy Pediatric Rehabilitation Gross Motor Function Range of Motion Gaza Strip
MeSH Terms: interventions — Myofascial Release Therapy

STUDY DESIGN:
Intervention Model Description: "Participants will be randomly assigned to one of two parallel groups: conventional physiotherapy only or conventional physiotherapy plus myofascial release."
Masking Description: "This is an open-label study; no masking of participants, care providers, investigators, or outcome assessors is implemented."
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Physiotherapy (CPT) (Active Comparator): "Participants will receive a standard conventional physiotherapy program following Achilles tendon surgery. The program includes stretching, strengthening, mobility, and functional training exercises designed to enhance recovery and improve lower limb function."
  Interventions: Other: Conventional Physiotherapy
- Conventional Physiotherapy + Myofascial Release (CPT + MFR) (Experimental): "Participants will receive the same conventional physiotherapy program as the control group combined with myofascial release technique. The manual therapy will be applied to the lower limb and ankle region to improve fascial mobility, enhance soft tissue flexibility, and increase ankle range of motion."
  Interventions: Other: Conventional Physiotherapy; Other: Myofascial Release Technique

INTERVENTIONS:
Other: Conventional Physiotherapy — A standard physiotherapy program provided after Achilles tendon surgery, including stretching, strengthening, mobility, and functional training exercises
Other: Myofascial Release Technique — A manual therapy technique applied to the lower limb and ankle region, aiming to release fascial restrictions, improve soft tissue flexibility, and enhance ankle range of motion.
  Arms: Conventional Physiotherapy + Myofascial Release (CPT + MFR)

SUMMARY:
"This study aims to evaluate the effectiveness of adding Myofascial Release (MFR) technique to a conventional physiotherapy program for children with cerebral palsy after Achilles tendon surgery. The primary goal is to determine whether MFR can improve functional outcomes such as gross motor function and ankle range of motion, compared to physiotherapy alone. The study will be conducted in Gaza, Palestine, with children diagnosed with cerebral palsy who recently underwent Achilles tendon surgery. Participants will be randomly assigned to either conventional physiotherapy or conventional physiotherapy combined with MFR, and outcomes will be assessed before and after an 8-week intervention program."

DETAILED DESCRIPTION:
"Children with cerebral palsy (CP) often develop musculoskeletal complications, including Achilles tendon contractures, which may require surgical intervention. Despite surgery, many children continue to experience limitations in functional mobility and reduced range of motion. Conventional physiotherapy programs are commonly provided postoperatively to enhance recovery; however, additional manual therapy techniques such as Myofascial Release (MFR) may further improve outcomes.

This randomized controlled trial investigates the effectiveness of adding MFR to conventional physiotherapy for children with CP after Achilles tendon surgery in Gaza. Participants will be randomly allocated to either a control group (conventional physiotherapy only) or an intervention group (conventional physiotherapy plus MFR). Functional outcomes, including gross motor function (GMFM-88) and ankle range of motion, will be measured pre- and post-intervention. It is hypothesized that children receiving MFR in addition to conventional physiotherapy will demonstrate greater improvements in functional mobility and ankle range of motion compared to those receiving physiotherapy alone."

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2-5 years
* Spastic cerebral palsy diagnosis (GMFCS levels I-IV).
* Underwent Achilles tendon surgery within the past 3 months
* Medically stable and cleared to begin physiotherapy.
* Parental/guardian consent to participate in the study.

Exclusion Criteria:

* Other neuromuscular disorders
* Severe cognitive impairments that hinder participation
* Previous MFR therapy within the last 6 months
* Participation in another rehabilitation study in the past 3 months.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-08-20 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Gross Motor Function Measure (GMFM-88) | Baseline and after 8 weeks of intervention
  Change in gross motor function measured using the GMFM-88 scale. The scale assesses motor function in children with cerebral palsy across five dimensions: lying & rolling, sitting, crawling & kneeling, standing, and walking/running/jumping. Higher scores indicate better motor function.

SECONDARY OUTCOMES:
Pediatric Balance Scale (PBS) | Baseline and after 8 weeks of intervention
  Change in balance performance measured using the Pediatric Balance Scale, which consists of 14 functional balance tasks. Higher scores indicate better balance ability.
Ankle Range of Motion (ROM) | Baseline and after 8 weeks of intervention
  Passive ankle dorsiflexion range of motion measured using a goniometer. Improved ROM indicates increased flexibility and joint mobility.

CONTACTS AND LOCATIONS:
Overall Officials: Ismail K Al Qedra, MSc (Physiotherapy), Principal Investigator — Al-Azhar University - Gaza; Musab M Al Dabbas, PhD, Study Director — Al-Azhar University - Gaza
Locations (1):
- The Jerusalem Princess Basma Centre - Al-Ahli Al-Arabi Hospital, Gaza, Gaza, Gaza Strip, Palestinian Territories

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the results reported in this article will be made available upon reasonable request from the Principal Investigator Ismail Kamal Al Qedra after publication. Data will be shared for academic and research purposes only.
Supporting Information: Study Protocol, SAP
Time Frame: IPD and supporting information will be available starting 6 months after publication of the primary results and for a period of 5 years thereafter.
Access Criteria: Access to de-identified IPD and supporting documents will be granted to qualified researchers upon reasonable request. Requests must include a methodologically sound proposal and will be reviewed by the Principal Investigator. Data will be shared via secure electronic transfer.

REFERENCES:
- [Background] Russell DJ, Rosenbaum PL, Avery LM, Lane M. Gross Motor Function Measure (GMFM-66 & GMFM-88) User's Manual. Cambridge University Press; 2002.
- [Background] Barnes MF. The basic science of myofascial release: morphologic change in connective tissue. J Bodyw Mov Ther. 1997;1(4):231-238.
- [Background] Novak I, Morgan C, Fahey M, Finch-Edmondson M, Galea C, Hines A, Langdon K, Namara MM, Paton MC, Popat H, Shore B, Khamis A, Stanton E, Finemore OP, Tricks A, Te Velde A, Dark L, Morton N, Badawi N. State of the Evidence Traffic Lights 2019: Systematic Review of Interventions for Preventing and Treating Children with Cerebral Palsy. Curr Neurol Neurosci Rep. 2020 Feb 21;20(2):3. doi: 10.1007/s11910-020-1022-z. PMID 32086598
- See also: ClinicalTrials.gov — https://www.clinicaltrials.gov

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-07-03): https://cdn.clinicaltrials.gov/large-docs/56/NCT07148856/Prot_SAP_000.pdf